CLINICAL TRIAL: NCT00633620
Title: Narrow Band Versus Conventional Endoscopic Imaging for Screening Colonoscopy in a Private Practice Setting - A Large Prospective Randomized Trial
Brief Title: Narrow Band Versus Conventional Endoscopic Imaging for Screening Colonoscopy
Acronym: BECOP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Thomas Rösch, M.D., Central Interdisciplinary Endoscopy Unit, Charité Berlin, CVK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Charite-CVK-Endo-1; Berlin Colonoscopy Project 2
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Adenoma
Keywords: colonoscopy; narrow band imaging; adenoma; diagnosis; colonoscopic adenoma detection
MeSH Terms: conditions — Adenoma; Disease | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- colonoscopy (Experimental): Non-NBI HDTV colonoscopy
  Interventions: Device: Olympus NBI colonoscope 180 HDTV narrow band imaging (diagnostic test)

INTERVENTIONS:
Device: Olympus NBI colonoscope 180 HDTV narrow band imaging (diagnostic test) — colonoscopy withdrawal with NBI mode
  Other Names: Olympus NBI colonoscope 180 HDTV

SUMMARY:
Narrow Band Imaging (NBI) with high-definition (HDTV) visualization has been implemented into GI endoscopy with the purpose to better highlight endoluminal pathological structures by improving their contrast. Previous studies from referral centers could not show significant differences in terms of colonoscopic adenoma detection rate, but either very high adenoma rates or some numerical differences suggested that some benefit may exist which may become evident with average adenoma rates and/or large case numbers.

In a prospective randomized trial performed exclusively in a multicenter private practice setting involving 6 examiners with substantial life-time experience (>10.000 colonoscopies) 1200 patients will undergo HDTV screening colonoscopy with either NBI or conventional imaging technique on instrument withdrawal. Primary outcome measure is the adenoma detection rate (ADR; i.e. number of adenomas per patient).

DETAILED DESCRIPTION:
in 5 private practices with 6 examiners, consecutive asymptomatic persons willing to undergo screening colonoscopy will be asked to participate in this randomized study.

After introduction of the colonoscope into the cecum, patients will be randomized into withdrawal with either the NBI mode or conventional imaging by using wide-angle colonoscopes with HDTV imaging (Olympus Corp., Hamburg, Germany) in both groups. Randomization lists will be used for group allocation in each individual practice. In the NBI group, switching back to conventional imaging, and the number of occasions for switching back and the reasons for it are documented in this group.

Patients bowel preparation consists mostly of polyethylene glycol lavage with 4-5 liters until clear rectal fluid is evacuated. All examiners shall take special care to wash and clean the entire large bowel during instrument introduction and withdrawal, in order to provide optimal imaging conditions.

The following parameters are documented:

* Age and sex of the patient
* Type and dosage of sedation
* Examination time, both for instrument introduction and withdrawal
* Polyp characteristics: size (measured by open forceps or snare), shape (pedunculated/elevated, sessile/flat, and location
* Polyp histology after removal using snare polypectomy or forceps removal (for polyps < 3 mm), or biopsy if there are contraindications
* Other lesions found such as cancers, diverticula, inflammatory lesions etc. The main outcome parameter is the adenoma detection rate (number of polyps/number of patients examined) in the two groups.

Secondary outcome measures include analysis of the total number of polyps, flat/sessile adenomas, small adenomas (< 1 cm), hyperplastic polyps with size determination and right-sided versus left-sided polyp location in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic persons > 55 years willing to undergo screening colonoscopy

Exclusion Criteria:

* Missing consent
* Symptomatic persons
* Poor general conditions, significant comorbidity

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1250 (Actual)
Dates: Start 2007-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate (number of polyps/number of patients examined) | 6 months

SECONDARY OUTCOMES:
analysis of the total number of polyps, flat/sessile adenomas, small adenomas (< 1 cm), hyperplastic polyps with size determination and right-sided versus left-sided polyp location | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. Dr., Principal Investigator — Charité Medical University Berlin
Locations (1):
- Charité University Hospitals, Campus Virchow Hospital, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Adler A, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Scheel M, Schroder A, Yenerim T, Wiedenmann B, Gauger U, Roll S, Rosch T. Latest generation, wide-angle, high-definition colonoscopes increase adenoma detection rate. Clin Gastroenterol Hepatol. 2012 Feb;10(2):155-9. doi: 10.1016/j.cgh.2011.10.026. Epub 2011 Nov 2. PMID 22056301
- [Derived] Adler A, Aschenbeck J, Yenerim T, Mayr M, Aminalai A, Drossel R, Schroder A, Scheel M, Wiedenmann B, Rosch T. Narrow-band versus white-light high definition television endoscopic imaging for screening colonoscopy: a prospective randomized trial. Gastroenterology. 2009 Feb;136(2):410-6.e1; quiz 715. doi: 10.1053/j.gastro.2008.10.022. Epub 2008 Oct 15. PMID 19014944